CLINICAL TRIAL: NCT05703646
Title: Safety and Clinical Performance of the Yukon Choice PC, Yukon Chrome PC & Yukon Choice Flex Sirolimus Eluting Bioabsorbable Polymer Stents Systems in Routine Clinical Practice: e-Yukon Global Registry.
Brief Title: Safety and Clinical Performance of the Yukon Choice PC, Yukon Chrome PC & Yukon Choice Flex Stents in Routine Practice
Acronym: e-Yukon
Status: Recruiting | Type: Observational
Sponsor: Translumina GmbH (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Other Study IDs: e-Yukon Global Registry
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Ischemic Heart Disease
Keywords: stent; ischemic heart disease; registry; international; routine practice
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to collect safety and performance information in the setting of a large-scale clinical registry.

Patients meeting the selection criteria will be included, in chronological order of their implantation. This registry does not require any additional procedures, follow-up interventions, or ionizing radiation for patients.

The inclusion period is planned to last 2 years, starting in Q1 2023. The study will be complete when data on all patient's follow-up for one year have been collected.

DETAILED DESCRIPTION:
* Prospective, observational, noninterventional, multicenter, international clinical registry
* Allocation: consecutively treated patients, non-randomized
* Masking: None (open label)
* Observational model: Longitudinal
* Inclusion period: 2 years
* Follow-up period: at 1 year
* Study duration: 3 years

Patients meeting the selection criteria will be included, in chronological order of their implantation. This registry does not require any additional procedures, follow-up interventions, or ionizing radiation for patients.

The inclusion period is planned to last 2 years, starting in Q1 2023. The study will be complete when data on all patient's follow-up for one year have been collected.

List of visits:

V0: During hospitalization: consultation baseline, data of the intervention and data at discharge

V1: consultation at 30 days Follow-Up

V2: consultation at 12 months Follow-Up

ELIGIBILITY:
Inclusion Criteria:

* Any patient who was implanted only with a Yukon Choice PC, a Yukon Chrome PC or/and a Yukon Choice Flex stent within previous 2 days.
* Patient ≥ 18 years old.
* Male or non-pregnant female patient (Note: females of childbearing potential must have a negative pregnancy test prior to enrollment in the study).

Exclusion Criteria:

* Currently enrolled in another investigational device or drug trial that has not completed the primary endpoint or that clinically interferes with the current study endpoints.
* Co-morbid condition(s) that could limit the patient's ability to participate in the trial or to comply with follow-up requirements or impact the scientific integrity of the trial.
* Concurrent medical condition with a life expectancy of less than 12 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with coronary artery lesions in native coronary arteries ranging from 2.00 mm to 4.00 mm
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure | 12 months
  Defined as the composite of cardiac death, target-vessel myocardial infarction and clinically indicated target lesion revascularization

SECONDARY OUTCOMES:
Device success | 12 months
  Defined as successful delivery and deployment of the assigned device at the intended target lesion and successful withdrawal of the delivery system with attainment of final in-stent residual stenosis of <30% (by visual estimation).
Procedure Success | 12 months
  Device success without the occurrence of an ischemia-driven major adverse cardiac event during the hospital stay to a maximum of first seven days post index procedure.
All cause death | 12 months
  Defined as the rate of death from any cause
Cardiac death | 12 months
  Defined as death resulting from cardiovascular causes
Myocardial infarction | 12 months
  Defined as the rate of myocardial infarction
Target-vessel myocardial infarction | 12 months
  Defined as a myocardial infarction occurring on the stented target vessel
Clinically driven target lesion revascularization | 12 months
  Defined as a repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication involving the target lesion
Any revascularization | 12 months
  defined as clinically driven target lesion revascularization or angiographically driven target lesion revascularization, performed due to angiographic detection of significant restenosis in a patient who is clinically asymptomatic.
Stent Thrombosis | 12 months
  Defined as a thrombotic occlusion of a coronary stent (definite or probable, as per Academic Research Consortium definitions)

CONTACTS AND LOCATIONS:
Overall Officials: ROBERT BYRNE, Professor, Principal Investigator — Cardiovascular Research RCSI University of Medicine and Health Sciences, Dublin, Ireland
Locations (1):
- Al Qassimi hospital, Sharjah city, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No